CLINICAL TRIAL: NCT06760078
Title: Safety and Efficacy of Intravenous Tranexamic Acid with Intensive Blood Pressure Management in Ultra-Early Intracerebral Hemorrhage
Brief Title: Tranexamic Acid with Intensive Blood Pressure Management in Ultra-Early Intracerebral Hemorrhage
Acronym: TIME-ICH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Municipal Health Commission (Other Government); Capital Medical University (Other); Suzhou First People's Hospital (Unknown); Linyi People's Hospital (Other); Peking University Care Luzhong Hospital (Other); Wuzhou Red Cross Hospital (Other); Yantai Penglai Traditional Chinese Medicine Hospital (Unknown); The First Affiliated Hospital of Hebei North University (Other); Jiaozuo Tumor Hospital (Unknown); Hunan Provincial People's Hospital (Other); The People's Hospital of Liaoning Province (Other); The First People's Hospital of Qujing, Yunnan Province (Unknown); Huizhou Third People's Hospital, Guangzhou Medical University (Other); Nanyang Nanshi Hospital, Henan University (Unknown); Xing'anmeng People's Hospital (Unknown); Beijing Aerospace Center Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIME-ICH
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Spontaneous Intracranial Hemorrhage; Hypertension
Keywords: Intracranial Hemorrhage; Tranexamic acid; Intensive blood pressure lowering; Haemostatic therapy
MeSH Terms: conditions — Hypertension; Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (TXA) group (Experimental): Intravenous tranexamic acid 1 g over 10 minutes, followed by 1 g over 8 hours, with intensive blood pressure lowering.
  Interventions: Drug: intravenous tranexamic acid (TXA) infusion
- Control group (Placebo Comparator): An intravenous placebo (normal saline) over 10 minutes, followed by another continuous infusion of placebo over 8 hours, with intensive blood pressure lowering maintained.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intravenous tranexamic acid (TXA) infusion — Intravenous tranexamic acid will be administered as an initial dose of 1 g (10mL: 1g, diluted in 90 mL normal saline) over 10 minutes, followed by a maintenance dose of 1 g over 8 hours (10mL: 1g, diluted in 240 mL normal saline). Intensive blood pressure lowering will be maintained throughout the treatment period until 24 hours after onset.
  Arms: Tranexamic acid (TXA) group
Drug: Placebo — An intravenous placebo (10mL NS, diluted in 90mL NS) matching the specification and appearance of TXA will be administered as an initial bolus over 10 minutes, followed by a continuous infusion of placebo (10mL NS, diluted in 240mL NS) over 8 hours, with intensive blood pressure lowering maintained throughout the treatment period and continued until 24 hours after symptoms onset.
  Arms: Control group

SUMMARY:
This is a prospective, multicenter, randomized, quadruple-blind, placebo-controlled study. This study aims to estimate the safety and efficacy of intravenous tranexamic acid (TXA) combined with intensive blood pressure lowering in ultra-early spontaneous intracerebral hemorrhage (ICH).

DETAILED DESCRIPTION:
This trial is designed to evaluate whether tranexamic acid can reduce hematoma expansion and improve functional outcomes when combined with intensive blood pressure lowering in cases of ultra-early intracerebral hemorrhage with a high risk of hematoma expansion.

Participants who meet the eligibility criteria will be randomly assigned in a 1:1 ratio to either the TXA therapy group or the placebo control group. The initial infusion of 1 g of TXA or a matching placebo, along with intensive blood pressure lowering treatment, should commence as quickly as possible, ideally within 30 minutes of randomization. Following this, an additional 1 gram of TXA or a corresponding placebo will be administered via continuous intravenous infusion over 8 hours. Both groups will receive intensive blood pressure management during the first 24 hours after the onset of symptoms. Participants will be followed for 90 days after randomization for efficacy and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years old;
2. A definite diagnosis of supratentorial brain parenchymal hemorrhage by non-contrast cranial CT scan;
3. Hemorrhage volume less than 40 mL, as calculated using the ABC/2 method, with ultra-early hemorrhage growth (uHG) 10 mL/h or higher;
4. A clear time of symptom onset, and the randomization must occur within 2 hours from the onset;
5. At least two measurements of systolic blood pressure that are ≥150 mmHg and <220 mmHg, with at least a 2-minute interval between measurements.;
6. Baseline NIHSS of 8 or higher, or unilateral limb muscle strength of 0-3 grades;
7. GCS score greater than 8;
8. The patient or their legal representative has signed an informed consent form.

Exclusion Criteria:

1. Pre-illness mRS > 2;
2. Primary thalamic hemorrhage or intracerebral hemorrhage that has extended into the ventricles;
3. Scheduled for surgical intervention (i.e., hematoma evacuation, craniectomy);
4. Secondary ICH from tumors, AVMs, and aneurysms;
5. Traumatic brain injury-related hemorrhage;
6. Recent stroke, TIA, or thrombolytic therapy;
7. On anticoagulants;
8. Blood disorders, platelets <50,000/µL, or INR ≥1.8;
9. Antihypertensive therapy contraindications;
10. Indications for immediate blood pressure reduction;
11. Active thrombosis or thromboembolic history;
12. Hereditary or acquired thrombophilia;
13. Acquired color vision deficiency;
14. Epilepsy history;
15. GFR <90 mL/min;
16. Elevated ALT or liver disease;
17. Allergy to TXA or antifibrinolytics;
18. Life expectancy <12 months;
19. Pregnant or lactating women;
20. In other interventional clinical trials;
21. Other investigator-defined ineligibilities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) of 0-3 at 90 days | 90 ± 7 days

SECONDARY OUTCOMES:
Hematoma expansion at 24 hours | 24±3 hours
  The expansion is defined as a 33% or 6 mL increase from baseline hematoma volume or develop an intraventricular hemorrhage.
Absolute intracerebral haematoma growth at 24 hours | 24±3 hours
Relative intracerebral haematoma growth at 24 hours | 24±3 hours
Intraventricular hematoma (IVH) growth at 24 hours | 24±3 hours
National Institutes of Health Stroke Scale (NIHSS) score at 24 hours | 24±3 hours
Neurologic deterioration in first 24 hours | 24±3 hours
  Neurologic deterioration is defined as an increase of 4 or more points on the National Institutes of Health Stroke Scale (NIHSS) from baseline to 24 hours, or a decline of 2 or more points on the Glasgow Coma Scale (GCS).
Received surgical intervention within 7 days | Within 7±3 days
  Interventions include hematoma evacuation, external ventricular drainage, and craniectomy.
modified Rankin Scale (mRS) score at 90 days | 90±7 days
modified Rankin Scale (mRS) score of 0-4 at 90 days | 90±7 days
Utility weighted modified Rankin Scale (mRS) score at 90 days | 90±7 days
Major thromboembolic events | Within 90±7 days
  This includes ischemic stroke, myocardial infarction, and pulmonary embolism.
Death due to any cause within 90 days | Within 90±7 days
Severe hypotension | Within 72 hours
  Hypotension with clinical consequences (including acute renal failure) that required corrective therapy with intravenous fluids, vasopressors, or hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhai Guo, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No